CLINICAL TRIAL: NCT02249026
Title: Sublingual Buprenorphine Treatment for Neonatal Abstinence Syndrome - Pilot Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gauda, Estelle B., M.D. (Individual)
Collaborators: Johns Hopkins University (Other); Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0501
Record Dates: First submitted 2014-08-11; First posted 2014-09-25 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Drug; Withdrawal Symptoms, Neonatal; Withdrawal; Fetus and Newborn Affected by Other Maternal Medication
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Buprenorphine, Naloxone Drug Combination; Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BZDs + opiate exposure treated with BPN (Experimental): In-utero opiate and BZD exposed neonates + Buprenorphine sub-lingual administered in dose volumes greater than 0.5 mL will be given in 2 aliquots separated by 2 minutes allowing time for the drug to be absorbed.
  Interventions: Drug: BZDs + opiate exposure treated with BPN
- Opiates exposure treated with BPN (Active Comparator): In-utero opiate exposed neonates + Buprenorphine sub-lingual administered in dose volumes greater than 0.5 mL will be given in 2 aliquots separated by 2 minutes allowing time for the drug to be absorbed.
  Interventions: Drug: Opiates exposure treated with BPN

INTERVENTIONS:
Drug: BZDs + opiate exposure treated with BPN — These infants will have been exposed not only to opiates but also to BZDs during pregnancy. Administration of Buprenorphine: The solution will be administered under the tongue followed by the insertion of a pacifier to reduce swallowing. Dose volumes greater than 0.5 mL will be given in 2 aliquots separated by 2 minutes allowing time for the drug to be absorbed. If the infant's withdrawal is not controlled, clonidine will be used as adjunct therapy. The initial dose of clonidine is 6 mcg/kg/day in 4 divided doses given every 6 hours. If signs of withdrawal are not controlled, the dose may be increased by 3mcg/kg/day to a maximum 12 mcg/kg/day divided q 6 hrs.
  Other Names: Suboxone; Subutex; Buprenex
  Arms: BZDs + opiate exposure treated with BPN
Drug: Opiates exposure treated with BPN — These infants will have been exposed not only to opiates during pregnancy. Administration of Buprenorphine: The solution will be administered under the tongue followed by the insertion of a pacifier to reduce swallowing. Dose volumes greater than 0.5 mL will be given in 2 aliquots separated by 2 minutes allowing time for the drug to be absorbed. If the infant's withdrawal is not controlled, clonidine will be used as adjunct therapy. The initial dose of clonidine is 6 mcg/kg/day in 4 divided doses given every 6 hours. If signs of withdrawal are not controlled, the dose may be increased by 3mcg/kg/day to a maximum 12 mcg/kg/day divided q 6 hrs.
  Other Names: Suboxone; Subutex; Buprenex
  Arms: Opiates exposure treated with BPN

SUMMARY:
Summary: There have been two published RCTs showing efficacy of buprenorphine treatment for NAS. However these trials excluded an estimated 22-47% of infants requiring pharmacologic treatment; those infants born to mothers with co-dependence on an opiate and a benzodiazepine. Although there are concerns, we anticipate that buprenorphine will be safe in this population. If it is safe, we can include these infants in the large double blind, double-dummy buprenorphine and clonidine vs. morphine and clonidine trial. If on the other hand, these infants have respiratory depression or other adverse events when buprenorphine is given, it will be important to report this study and caution the use of buprenorphine in these infants

DETAILED DESCRIPTION:
The Problem: Infants who are born to mothers taking or abusing opiates frequently suffer from neonatal abstinence syndrome (NAS) after birth. They often have withdrawal symptoms which can be life threatening if untreated. The American Academy of Pediatrics recommends opioid replacement for the treatment of these symptoms in newborns. Buprenorphine (BNP) has gained widespread use in the treatment of adult opioid dependence. One of the reasons BNP is so appealing is because of its safety profile in comparison to the other drugs in its class (opiates). It has less respiratory depression and a lower level of physical dependence than the other opioids. BNP has recently been trialed, in its sublingual form, as a treatment for newborns with NAS. In two trials by the same group, there was a significant reduction in both the length of treatment and in-patient hospital days in infants treated with BNP in comparison to infants treated with morphine.

In both of these studies, mother/infant pairs were excluded if the mother was dual dependent on opiates and benzodiazepines (BZDs). This is not an insignificant population. BZDs are frequently prescribed during pregnancy to treat anxiety and panic disorder in women who are taking methadone or BNP for opioid replacement therapy. BZDs are also common drugs of abuse. It has been estimated that 22-47% of mothers whose infants are diagnosed with NAS used both BZDs and opiates during the pregnancy. These infants have a protracted NAS with longer hospitalization in comparison to infants exposed to an opioid alone. There are conflicting reports in the literature regarding the safety of concomitant use of BNP and BZDs. In both adults and children the combination of BNP and BZD prolongs respiratory depression in non-drug abusers. In addition, autopsy findings in six adults who were drug abusers were linked to concomitant use of BNP and BZD by analysis at autopsy. On the other hand in adult tapering trials comparing BNP with methadone in dual-dependent adults there were no adverse events in the BNP group, opiate withdrawal scores were lower and the adults were more likely to complete treatment. Thus while treatment of NAS with BNP may be desirable and efficacious in opiate tapering protocols, it is imperative that we look specifically at this group of infants with dual exposure to opioids and BZDs. This is a single site, un-blinded observational safety study. Study participants will be recruited from eligible participants who are born at Bayfront Medical Center Baby Place and subsequently admitted to the neonatal intensive care unit (NICU) at All Children's' Hospital (ACH) for treatment of NAS. Data from this pilot safety trial will be used to apply for NIH funding to conduct a large randomized double-blind trial to determine the efficacy of BNP versus morphine for the treatment of NAS.

The Research Hypothesis: BNP can be used safely to treat NAS in the subgroup of infants whose mothers were taking both an opiate and a BZD in the week prior to delivery.

The Importance of the Research: BNP is emerging as a "safer" and more efficient drug for adult detoxification and maintenance programs and is showing promise for the treatment of neonatal abstinence syndrome (NAS). In the most recent published trial comparing BNP to morphine in infants with NAS, the length of stay (LOS) was decreased by 40% in the BNP group (from an average of 38 days in the morphine group to 23 days in the BNP group). No major adverse effects were reported in either treatment group. As is common in early trials, the experimental group was restricted - specifically maternal BZD use was an exclusion criteria. The rational given was that length of stay is known to be longer for infants whose mothers were also using BZDs. However, this is not an insignificant population. It has been reported that 22-47% of opiate users are co-using BZDs. At ACH, the incidence of infants exposed to both classes of drugs has ranged from 15-35%. Before BNP becomes the standard of care it is important to look closely at this group of infants and either caution the use of BNP or demonstrate its safety. This pilot trial is designed to determine if infants who have dual in-utero exposures to opiates and BZDs can be safely treated with BNP.

ELIGIBILITY:
Inclusion Criteria:

* Newborns ≥ 35 0/7 wks. Gestation undelivered or < 12 hours of age at enrollment and within the 72 hrs. after birth at the time of transfer to ACH for pharmacologic treatment for moderate to severe NAS
* Newborns ≥ 2 kg weight at birth (10th % for a 35 0/7 wk. newborn)
* Informed parental

Exclusion Criteria:

* Newborns <35 0/7 wks. gestation OR older than 72 hrs. of life at time of transfer to ACH for pharmacologic treatment for moderate to severe NAS
* Major congenital anomalies
* Major concomitant medical illness including antibiotic treatment for greater than 3 days
* Any illness that precludes oral or sublingual medication use
* Infants who have received any drug other than "study drug" to treat their NAS
* Infants requiring drug therapy with any high or moderate CYP3A4 inhibitor or inducer (Appendix A)
* Breastfeeding infants.
* Infants in significant pain requiring medication for comfort (for example those with a fracture).

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of vital signs | 2-8 weeks
  To determine the in infants with NAS who have in-utero exposure to opiates and BZDs. This is an un-blinded observational safety study. A total of 24 neonates with moderate to severe NAS will be enrolled at ACH and its obstetric affiliate Bayfront Hospital in Florida. 12 of these infants will have a positive screen (described below) for both maternally transferred opiate and BZD. The comparison group of 12 infants will have been exposed to opiates but not to BZDs during the pregnancy. Comparisons will be made both within and between groups. The principle outcome measures will be 1) respiratory function as measured by respiratory rate 2) a combined event score which includes episodes of apnea (>20 sec apneic pause), bradycardia (<80 bpm) and oxygen hemoglobin desaturation measured by pulse oximetry (<90%).
  Other safety measures will include: blood pressures.

SECONDARY OUTCOMES:
To determine BNP levels in blood, urine, and meconium(stool) | 2 - 8 weeks
  Secondary Objectives: To gain additional knowledge about the pharmacokinetics and pharmacodynamics of BNP and BZD in these neonates. Infant blood, urine, and meconium(stool) samples will be analyzed by mass spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle B Gauda, MD, Principal Investigator — JHMI
Locations (1):
- All Children's Hopsital, St. Petersburg, Florida, United States